CLINICAL TRIAL: NCT01367717
Title: Effect of Creatine Monohydrate and Creatine Ethyl Ester on Serum and Urinary Creatinine
Brief Title: Effect of Creatine on Serum and Urine Creatinine
Acronym: ECSUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 034-09
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Acute Kidney Injury
Keywords: Creatine; Creatinine; Serum Creatinine; Urine Creatinine; Creatine Monohydrate; Creatine Ethyl Ester; Acute Kidney Injury; Renal; Kidney
MeSH Terms: conditions — Acute Kidney Injury | interventions — Creatine; creatine ethyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Creatine Monohydrate (Active Comparator): Each of the 25 subjects took Creatine Monohydrate.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Creatine Ethyl Ester (Active Comparator): Each of the 25 subjects took Creatine Ethyl Ester.
  Interventions: Dietary Supplement: Creatine Ethyl Ester

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Each subject ingested 10 grams of commercially available creatine monohydrate orally. This was equivalent to two teaspoons according to the manufacturer's recommendations. The creatine was then solubilized in 8 oz. of water and 2 tablespoons of Tang brand orange flavored drink mix.
  Other Names: GNC Pro Performance Fruit Punch Creatine Monohydrate; Tang brand Orange Drink, manufactured by Kraft Foods
  Arms: Creatine Monohydrate
Dietary Supplement: Creatine Ethyl Ester — Each subject ingested 10 grams of creatine ethyl ester orally. This was equivalent to 14.25 pills according to the manufacturer's ingredient description. The pill capsules were ground into a powder, which was added to 8 oz of water along with 2 tablespoons of Tang brand orange drink.
  Other Names: CE2 Rapid Absorption Ester Creatine: Platinum; Tang brand Orange Drink, manufactured by Kraft Foods
  Arms: Creatine Ethyl Ester

SUMMARY:
Background: Creatinine (Crn) concentration is used to assess renal function via calculation of GFR (Glomerular Filtration Rate). By RIFLE (Risk, Injury, Failure, Loss, End Stage Kidney Disease) criteria, acute kidney injury (AKI) and acute renal failure (ARF) are defined by a two-fold and three-fold increase in serum Crn, respectively. Crn is a breakdown product of proteins and circulating creatine, and it is generally a benign product present in serum. Creatine is a nutritional supplement that has been available since 1993, and it is widely used among athletes today.

Methods: In an IRB approved, blinded crossover trial, 25 human volunteers ingested 2 creatine supplements to determine any associated statistically significant increase in serum Crn and clinically significant increase in serum Crn to a degree associated with AKI or ARF. Urine samples were also collected to examine excretion patterns after an ingested sample. Participants ingested 10 gm of creatine ethyl ester (CEE) or creatine monohydrate (CrM) and had serum Crn assayed at 0, 1, 2, 3, 4, 5 and 24 hours. Urinary Crn levels were assayed at 0, 1.5, 3, 5 and 24 hours. Exclusion factors were any history of renal disease or use of creatine within the last month. Statistical analysis was performed by Wilcoxon Matched-Pair Signed Ranks Test and descriptive summary statistics were performed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Human

Exclusion Criteria:

* Use of any form of creatine within 4 weeks prior to participation in study.
* Pregnancy
* History of elevated creatinine or renal insufficiency
* History of PKU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Serum Creatinine | 24 Hours
  Participants ingested 10 grams of creatine monohydrate or creatine ester and had serum creatinine measured at 0, 1, 2, 3, 4, 5, and 24 hours.
Urine Creatinine | 24 hours
  Participants ingested 10 grams of creatine monohydrate or creatine ethyl ester and had urinary creatinine levels measured at 0, 1.5, 3, 5, and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher K Hunt, M.D., Principal Investigator — Beth Israel Medical Center; Robert J Hoffman, M.D., Study Director — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States